CLINICAL TRIAL: NCT02938455
Title: Explorative Study About the Degree of DNA Methylation Related to Acute Perioperative Pain Treatment
Brief Title: DNA Methylation and Perioperative Pain Treatment
Acronym: MEDAPO
Status: Completed | Type: Observational
Sponsor: University of Bologna (Other)
Responsible Party: Principal Investigator, Andrea Fanelli, MD, University of Bologna
Other Study IDs: MEDAPO
Record Dates: First submitted 2016-10-17; First posted 2016-10-19 (Estimated); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Hyperalgesia; Pain, Postoperative
Keywords: Hyperalgesia; Opioids; Postoperative pain; DNA methylation
MeSH Terms: conditions — Hyperalgesia; Pain, Postoperative

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: No

SUMMARY:
In the last few years much attention has been paid to hyperalgesia induced by opioids, which represents a clinically significant condition following acute and chronic exposure to opioids. It has been suggested that the increase in gene expression of μ-opioid receptors and the development of hyperalgesia could be linked to epigenetic mechanisms. In particular the use of opioids seems to be related to an increase of the degree of DNA methylation. In the literature are not currently available data about the degree of DNA methylation in surgical patients, opioid-naive prior to surgery, receiving acute opioids treatment in the perioperative period.

The primary objective of this study is to assess the degree of perioperative DNA methylation (extracted from whole blood) in patients undergoing major surgery exposed to opioids according to current clinical practice compared to preoperative baseline levels. The timing (preoperative vs intraoperative vs postoperative) in which the possible increase of the degree of DNA methylation will happen wil be assessed.

20 consecutive patients undergoing major surgery performed under general anesthesia that have expressed their consent to participate to the study will be enrolled. This sample is adequate to allow the observation of a possible increase of DNA methylation in opioid-naive patients exposed to anesthesia/analgesia based on opiates according to current clinical practice.

DETAILED DESCRIPTION:
During perioperative period surgical patients experience profound changes in their physiological processes. In addition to surgical stress, these variations are in part due to pharmacological treatments commonly used for anesthesia and analgesia during and after surgical procedure.

Opioids are essential drugs for the management of acute perioperative pain. In the last few years much attention has been paid to hyperalgesia induced by opioids, which represents a clinically significant condition following acute and chronic exposure to opioids. It has been suggested that the increase in gene expression of μ-opioid receptors and the development of hyperalgesia could be linked to epigenetic mechanisms.

Epigenetic alterations typically involve changes in chromatin structure, which is composed of DNA, histones and non-histone proteins. Main changes in clinical setting are covalent modifications of N-terminal sequences of histone proteins and DNA methylation. In particular, DNA methylation is carried out with the addition of a methyl group on the fifth carbon atom of cytosine residues (5mC), mainly localized in CpG regions.

DNA methylation is considered as a mechanism of gene silencing. It is a complex process regulated by a whole family of enzymes called DNA methyl-transferase (DNMTs: DNMT1, DNMT2, DNMT3a, DNMT3B, and DNMT3L) that catalyze the transfer of a methyl group.

In particular DNMT 1, 3a, 3b were studied during the development of a neuropathic pain model. Through immunohistochemical analysis it was observed that in the dorsal root ganglion of an adult rat (L4-5) DNMT3B showed an important up-regulation that is observed already 1 week after the induction of the model and that persists for 4 weeks; on the contrary, DNMT1 and DNMT3a showed a moderate and transient up-regulation. Other studies have shown that in a different pattern of pain, acute inflammatory, the expression levels of DNMT3a and DNMT3B are particularly high.

All these findings suggest the important activity of these enzymes in different models of pain.

Opioids admnistration seems to be related to an increase of the degree of DNA methylation. In a study published in 2013, Doehring et al. rated the degree of DNA methylation in patients heroin addicts undergoing methadone substitution treatment. Patients treated with opioids have shown an overall increase in DNA methylation, in particular of μ-opioid receptor. It is interesting to note that the degree of DNA methylation correlates with the intensity of pain reported by subjects analyzed in the study.

In the literature are not currently present data related to the degree of DNA methylation in surgical patients receiving acute treatment with opiates that are opioid-naive prior to surgery.

The primary objective of this study is to assess the degree of perioperative DNA methylation (extracted from whole blood) in patients undergoing major surgery exposed to opiates according to current clinical practice compared to preoperative baseline levels. The timing (preoperative vs intraoperative vs postoperative) in which the possible increase of the degree of DNA methylation will happen will be assessed.

The secondary objectives are: observe the possible correlation between the degree of DNA methylation and the intensity of acute postoperative pain, observe the possible correlation between the degree of DNA methylation and the incidence of postoperative nausea and vomiting, observe the possible correlations between the degree of DNA methylation and the gene expression of μ opioid receptor, observe the possible correlations between the degree of DNA methylation and the expression of genes mainly involved in methylation processes, compare the degree of DNA methylation in the preoperative phase of the different patients involved in the study.

MEDAPO trial is a monocentric clinical trials with the use of human tissue in vitro. Because the lack of knowledge in literature about the increased degree of DNA methylation following acute administration of opioids in surgical patients, this study will be explorative. Moreover, not being able to avoid exposure to opiates in the intraoperative phase, but being possible to guarantee postoperative analgesia without opioid treatments, it will be interesting to see if any increase in methylation occurs already during the intraoperative phase or whether it can be related to the time of exposure to treatment with opiates.

This will provide useful information to better plan the timing for randomization into a future trial comparing various postoperative analgesic techniques.

20 consecutive patients undergoing major surgery performed under general anesthesia that have expressed their consent to participate to the study will be enrolled. This sample is adequate to allow the observation of a possible increase of DNA methylation in opioid-naive patients exposed to anesthesia/analgesia based on opiates according to current clinical practice.

Descriptive analysis related to the primary objective of the trial will be performed. We will perform parametric tests for paired data to observe the correlation between the degree of DNA methylation and acute postoperative pain.

After verifying the signature of informed consent, the presence of the inclusion criteria and the absence of exclusion criteria, the patient will be considered eligible. Each patient will be assigned to a serial number which will identify the samples used for molecular analysis making them anonymous.

The study period will extend from the signing of informed consent up to 48 hours after the end of surgical procedure.

The participation to the study will not change the treatment plan of the patient: surgical procedure and anesthetic conduct will represent the normal daily clinical practice without any variation regardless the enrollment of the patient.

At the time of arrival in the operating room the patient will be monitored according to standard clinical practice in relation to the type of surgery (ECG, SpO2, EtCO2 and Invasive Blood Pressure). After monitoring the patient, it will be placed a peripheral venous catheter ≤ 20 G and an arterial catheter (20G) in radial or humeral artery.

After adequate oxygenation anesthesia will be induced with fentanyl (3 mcg/kg), propofol (2-2.5 mg/kg) and Rocuronium (0.6 mg/kg) or Succinylcholine (1 mg/Kg). The maintenance of anesthetic level will be obtained by the use of Sevoflurane 0.7 - 1.3 MAC (minimum alveolar concentration), and bolus doses of Fentanyl (1mcg /kg) and possibly of Rocuronium (0.15mg/kg) every 45 minutes until the end of surgery.

The acute postoperative pain in the first 48 hours will be treated with a continuous intravenous infusion of morphine (1 mg/h), with the possibility of the patient to self-administer boluses of 1 mg of morphine repeatable every 8 minutes.

Continuous infusion of morphine will be preceded by an intraoperative bolus (immediately after the last stitch) of 0.1 mg/kg of morphine. Ten minutes after awakening the patient, if the pain will be poorly controlled (NRS ≥ 4), will be administered 1 mg of morphine, repeatable every 5 minutes, until NRS<3.

Prophylaxis for postoperative nausea and vomiting will carried out by intravenous administration of 0.1 mg/kg of dexamethasone prior to administration of the first dose of fentanyl. In case of postoperative nausea and vomiting, it will be administered droperidol 0.625 mg repeatable every 6 hours.

During the study period, in addition to the anthropometric parameters, we will collect the following data:

Duration of anesthesia, defined as the time between induction of general anesthesia and awakening; Duration of surgery, defined as the time between surgical incision and the last stitch; Fentanyl consumption, expressed in mcg/kg /hour; Morphine consumption in the first 24 and 48 hours after the end of surgery; Pain (NRS) at rest and after deep inhalation 10 minutes after waking up, 24 and 48 hours after the end of surgery; Number of episodes of nausea and vomiting in the first 24 and 48 hours after the end of surgery; Consumption of antiemetic drugs in the first 24 and 48 hours after the end of surgery.

During the study period, in addiction to blood tests carried out according to routine clinical practice a blood sample of 5 ml will be collected to perform epigenetic analysis. The semple will be added with heparin or EDTA or ascorbate ACD as anticoagulant agents and stored at a temperature of - 20 ° C until the delivery to the Department of Pharmacy and Biotechnology which will take place after the last blood sampling.

Samples will be collected according to the following schedule reflects everyday clinical practice:

* T0: after placement of the arterial catheter, prior to administration of opiates (baseline blood gases);
* T1: 1 hour after general anesthesia induction (hemogasanalysis verification of mechanical ventilation);
* T2: after the last stitch, before the intraoperative bolus of morphine (hemogasanalysis testing blood loss);
* T3: 24 ± 6 hours after after the end of surgery (control blood count);
* T4: 48 ± 6 hours after the end of surgery (control blood count). On these blood samples, it will be assessed the degree of DNA methylation. The samples will be subjected to extraction of RNA and genomic DNA through ZR-Duet ™ kit DNA / RNA Miniprep (Zymo Research). The nucleic acids obtained from the samples will be stored at - 80 ° C until analysis.

Since the change in methylation of genomic DNA is observed in various diseases, the need to measure the degree of overall DNA methylation has become very important. The 5-mC DNA ELISA kit (Zymo Research) offers a method of high-throughput, easy to identify and quantify the degree of DNA methylation.

Total RNA extracted from each sample will be used for gene expression studies using RT-qPCR method. This technique will allow making a quantitative assessment of genes' expression codifying for the μ opioid receptor and enzymes belonging to the family of DNMTs. Based on these results, we will be able to correlate the degree of DNA methylation to the levels of expression of the investigated genes.

ELIGIBILITY:
Inclusio Criteria: patients schedule for major surgery (longer than 120 minutes) exposed to opioid in the perioperative period; patients opioid naive prior to surgery; ASA < 4; 17 < BMI < 36.

Exclusion Criteria: renal and hepatic failure; OSAS; Apfel score > 3.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient undergoing elective major surgery under general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2016-10; Primary Completion 2020-05 (Actual); Study Completion 2020-05 (Actual)

PRIMARY OUTCOMES:
DNA Methylation | 2 days

CONTACTS AND LOCATIONS:
Locations (1):
- Andrea Fanelli, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No